CLINICAL TRIAL: NCT06763796
Title: Postural Decoding Technique for Treating Post-Stroke Shoulder Pain: A Clinical Randomized Controlled Trial.
Brief Title: Postural Decoding for Post-Stroke Shoulder Pain: A RCT.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Baoan District Fuyong People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2024-90; 2024JD056 (Other Grant/Funding Number: Shenzhen Bao'an District Science and Technology Bureau.)
Record Dates: First submitted 2025-01-01; First posted 2025-01-08 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Sequelae
Keywords: Hemiplegic Shoulder Pain；Postural Decryption Technique；Musculoskeletal Ultrasound Assessment；Postural Assessment； Randomized Controlled Trial
MeSH Terms: conditions — Stroke | interventions — Medicine, Chinese Traditional; Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Postural Decryption Technique Group) (Active Comparator): Assessment:
  PDT begins with visual inspection and palpation to assess neutral alignment of the trunk, spine, and shoulder complex. Evaluations proceed distal to proximal through coronal, sagittal, and transverse planes, focusing on joint symmetry.
  Treatment:
  The 4R Technique includes:
  1. Reposition - Correct joint alignment.
  2. Restore - Release soft tissue adhesions.
  3. Reinforce - Strengthen stabilizing muscles.
  4. Retrain - Improve movement patterns.
  Key Steps:
  1. Lumbar and Thoracic Adjustments: Manual traction, side-bending, and mobilizations.
  2. Scapular Realignment: Mobilization and muscle stretching.
  3. Joint Mobilization: Multi-directional gliding within pain-free ranges.
  4. Trigger Point Release: Pressure therapy for 5-10 seconds to relieve pain.
  Treatment Plan:
  4 weeks, 5 sessions per week, 40 minutes per session. Targets pain relief, range of motion, and postural correction in hemiplegic shoulder pain (HSP) patients.
  Interventions: Other: Postural Decryption Technique
- Control Group: Traditional Massage Group (Active Comparator): Treatment:
  The control group receives traditional massage therapy focused on:
  1. Soft Tissue Relaxation - Kneading, pressing, and rolling to reduce muscle tension.
  2. Joint Mobilization - Passive movements to improve range of motion (ROM). Pain Relief Techniques - Acupressure and trigger point therapy to ease pain and spasms.
  Treatment Plan:
  4 weeks, 5 sessions per week, 40 minutes per session. Targets pain relief, ROM improvement, and muscle relaxation in hemiplegic shoulder pain (HSP) patients.
  Interventions: Other: Traditional Chinese Medicine (TCM) Massage Therapy

INTERVENTIONS:
Other: Postural Decryption Technique — Assessment:
  PDT begins with visual inspection and palpation to check postural alignment and identify joint or muscle imbalances. Evaluations proceed distal to proximal, examining the spine and shoulder complex in coronal, sagittal, and transverse planes to assess symmetry and neutral positioning.
  Treatment Process:
  PDT applies the 4R Technique:
  1. Reposition - Correct joint alignment.
  2. Restore - Release muscle tension and adhesions.
  3. Reinforce - Strengthen stabilizing muscles.
  4. Retrain - Improve movement patterns and posture.
  Key Techniques:
  1. Spinal and Shoulder Adjustments: Manual traction, mobilizations, and stretches.
  2. Joint Mobilization: Multi-directional gliding within pain-free ranges.
  3. Trigger Point Therapy: 5-10 seconds of pressure to relieve localized pain.
  4. Proprioception Training: Balance challenges to improve stability and control.
  Arms: Intervention Group (Postural Decryption Technique Group)
Other: Traditional Chinese Medicine (TCM) Massage Therapy — Definition:
  A manual therapy based on Traditional Chinese Medicine (TCM) principles, using techniques like kneading, pressing, rolling, and stretching to relieve pain, improve circulation, and enhance mobility.
  Key Features:
  1. Techniques: Soft tissue manipulation, joint mobilization, and acupressure.
  2. Focus: Pain relief, joint function recovery, and muscle relaxation.
  Treatment Plan:
  4 weeks, 5 sessions per week, 40 minutes per session.
  Arms: Control Group: Traditional Massage Group

SUMMARY:
Brief Summary

Purpose of the Study:

This clinical trial aims to determine whether Postural Decryption Technique can effectively treat hemiplegic shoulder pain (HSP) in patients recovering from stroke. It also seeks to assess the safety of this technique. The study will compare the effectiveness of the Postural Decryption Technique with traditional massage therapy to find out which method provides better pain relief and improves shoulder function.

Key Research Questions:

1. Can the Postural Decryption Technique reduce shoulder pain and improve range of motion in HSP patients?
2. Is the Postural Decryption Technique more effective than traditional massage therapy?
3. Is the Postural Decryption Technique safe, and are there any side effects or discomfort during treatment?

   Study Design:
4. Researchers will recruit 48 participants with HSP and randomly divide them into two groups:

Treatment Group: Participants will receive therapy using the Postural Decryption Technique.

Control Group: Participants will undergo traditional massage therapy.

What Participants Will Do:

Receive treatment 5 times per week, 40 minutes per session, for 4 weeks. Undergo evaluations before treatment, 2 weeks after treatment begins, and at the end of 4 weeks to measure pain relief and shoulder function improvement.

Undergo musculoskeletal ultrasound to assess changes in soft tissue and joint structure.

Evaluation Methods:

1. Pain Assessment: Pain levels will be measured using the Visual Analog Scale (VAS).
2. Range of Motion (ROM): Tools will be used to measure the angles of shoulder movement.
3. Postural Assessment: The position of the scapula and spine will be measured to evaluate postural alignment improvements.
4. Daily Activity Ability: Progress in daily tasks will be recorded using the Barthel Index questionnaire.

Significance of the Study:

This study aims to validate whether the Postural Decryption Technique is a more effective and safer treatment for HSP compared to traditional massage therapy. If proven effective, it could offer a new rehabilitation approach to reduce pain, restore function, and improve the quality of life for stroke survivors.

Safety Monitoring:

Researchers will closely monitor participants for any signs of discomfort or adverse effects during the treatment process. Participants are free to withdraw from the study at any time if they experience any issues.

Conclusion:

The ultimate goal of this study is to identify a better treatment option for HSP in stroke patients. The results are expected to support the application of the Postural Decryption Technique as a safe and effective rehabilitation method for broader clinical use.

DETAILED DESCRIPTION:
Section 1: Introduction to Postural Decryption Technique (PDT)

Background and Development:

The Postural Decryption Technique (PDT) was co-developed by Professor Won Sang-Hee from South Korea and Professor Wang Qiang from the Rehabilitation Medicine Department of the Affiliated Hospital of Qingdao University. This innovative rehabilitation approach integrates biomechanical assessments with precise interventions to correct joint alignment, restore muscle function, and retrain movement patterns.

Professor Wang Qiang has dedicated years to applying PDT for the treatment of shoulder joint adhesions and gait dysfunctions in patients with hemiplegic shoulder pain (HSP) after stroke. His work has demonstrated remarkable clinical efficacy and laid a solid foundation for the broader application of this technique in rehabilitation medicine.

Core Principles and Technical Framework:

PDT emphasizes the importance of postural alignment and joint stability in rehabilitation. It is based on the 4R Core Technique, which includes:

1. Reposition - Correcting abnormal joint alignments to restore normal positioning and stability.
2. Restore - Releasing soft tissue adhesions to improve muscle elasticity and flexibility.
3. Reinforce - Strengthening key muscle groups and enhancing neuromuscular control.
4. Retrain - Re-educating patients in functional movements to maintain proper posture and prevent recurrence.

Features and Advantages:

1. Addresses Root Causes: Unlike conventional treatments that focus on symptom relief, PDT targets the biomechanical imbalances that lead to pain and dysfunction.
2. Personalized Approach: Treatment plans are customized based on individual postural assessments and functional limitations, ensuring optimal outcomes.

   Non-Invasive Therapy: PDT is safe, painless, and well-tolerated, making it suitable for long-term application.
3. Broad Applicability: Beyond treating HSP, PDT has shown positive results in managing chronic pain, gait impairments, and spinal deformities such as scoliosis.

Section 2: Study Design

Study Framework:

This study adopts a randomized controlled trial (RCT) design to evaluate the clinical efficacy and safety of PDT in treating HSP. It also compares PDT with traditional massage therapy to determine the superior approach.

Participants:

A total of 48 eligible participants diagnosed with HSP will be randomly assigned into two groups:

PDT Group (Treatment Group): Participants will undergo therapy using the Postural Decryption Technique.

Traditional Massage Group (Control Group): Participants will receive standard massage therapy.

Intervention Methods:

Postural Decryption Technique (PDT Group):

Evaluation: Analyze scapular alignment, thoracic posture, and joint biomechanics to identify dysfunctions.

4R Protocol: Apply repositioning, soft tissue release, muscle reinforcement, and movement retraining.

Focus Areas:

Joint Mobilization: Sliding and stretching of the glenohumeral joint to improve range of motion.

Muscle Relaxation: Release tight muscles (e.g., pectoralis minor, serratus anterior).

Scapular Stabilization: Proprioception exercises to enhance balance and neuromuscular control.

Functional Retraining: Teach proper movement patterns to maintain postural alignment.

Traditional Massage Therapy (Control Group):

Soft tissue relaxation techniques (kneading, pressing). Passive joint mobilization for improved flexibility. Pain relief methods, such as acupressure and trigger point therapy.

Treatment Duration:

5 sessions per week, 40 minutes per session, for 4 weeks. Adjustments to intensity and methods will be made based on participant progress.

Outcome Assessments:

Primary Outcomes:

Pain Relief (VAS): Visual Analog Scale (0-10) to measure pain intensity. Range of Motion (ROM): Goniometer to assess flexion, abduction, and extension angles.

Secondary Outcomes:

Functional Independence (Barthel Index): Measures daily activity performance, scored 0-100.

Postural Symmetry: Vertical distance between scapular angles and the second thoracic vertebra, evaluated for alignment improvement.

Musculoskeletal Ultrasound: Tracks changes in muscle structure, tendon thickness, and joint effusion.

Safety Monitoring:

Record adverse events, such as increased pain, swelling, or loss of function. Allow participants to withdraw at any stage if discomfort occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for stroke.
2. Presence of stroke-related lesions confirmed by cranial CT or MRI.
3. Hemiplegic shoulder pain and motor dysfunction on the affected side.
4. Shoulder pain occurring after paralysis, with a VAS score ≥ 5.
5. ≥ 18 years.
6. First-ever stroke, presenting with unilateral limb paralysis, and classified
7. between Stages II-V based on Brunnstrom motor function recovery stages.
8. No severe cognitive impairment, with normal cognitive function assessment. Signed informed consent form.

Exclusion Criteria:

1. Subarachnoid hemorrhage.
2. History of two or more strokes.
3. Shoulder subluxation in the flaccid stage.
4. Disease progression with new infarction or hemorrhagic lesions.
5. Severe cardiopulmonary diseases, including acute myocardial infarction, unstable angina, myocardial ischemia detected on resting ECG, severe arrhythmias, aortic stenosis, acute pericarditis, or malignant hypertension.
6. Shoulder pain caused by cervical spondylosis, periarthritis, sports injuries, gallbladder disease, thalamic lesions, or myocardial infarction.
7. Severe psychological or cognitive impairments that prevent cooperation with treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
VAS（Visual Analog Scale） | The assessment time points are before treatment, 2 weeks after treatment, and 4 weeks after treatment.
  In the Visual Analog Scale (VAS) scoring system, patients are presented with an unmarked line that is 10 centimeters long. Patients indicate their level of pain by marking a point along the line. The position of the mark is measured using a ruler, yielding a corresponding numerical value. The VAS score ranges from 0 to 10, where 0 represents no pain and 10 represents the most severe pain. Higher scores indicate greater pain intensity.
Range of motion，ROM | The assessment time points are before treatment, 2 weeks after treatment, and 4 weeks after treatment.
  A goniometer is used to measure the flexion, abduction, and extension range of motion (ROM) of the shoulder joint in both groups of patients.
The absolute value of the vertical distance difference between the medial superior angle of the scapula on the affected side and the spinous process of the second thoracic vertebra (T2). | The assessment time points are before treatment, 2 weeks after treatment, and 4 weeks after treatment.
  The patient sits comfortably with arms relaxed at their sides. The medial superior angle of the scapula is marked as Point 1, and the spinous process of the second thoracic vertebra (T2) is marked as Point 2. A ruler or measuring tape is used to measure the vertical distance between these two points. The absolute value of the distance difference before and after treatment is recorded to evaluate the effectiveness of the intervention, with a smaller difference indicating improved scapular alignment and postural symmetry.

SECONDARY OUTCOMES:
Barthel Index | The assessment time points are before treatment, 2 weeks after treatment, and 4 weeks after treatment.
  The Barthel Index is an assessment tool used to evaluate a patient's ability to perform activities of daily living (ADLs). It includes tasks such as eating, bathing, and dressing, with each activity scored based on the patient's level of independence. Higher scores indicate greater functional independence, while lower scores reflect a greater need for assistance.
musculoskeletal ultrasound | The assessment time points are before treatment, 2 weeks after treatment, and 4 weeks after treatment.
  Musculoskeletal ultrasound is an effective method for evaluating soft tissue abnormalities around the shoulder joint, offering high sensitivity and accuracy. It plays a crucial role in the clinical diagnosis and treatment of shoulder disorders. During the ultrasound examination, two musculoskeletal ultrasound specialists independently scan each patient using a blinded method. If their findings are consistent, the result is confirmed. If there is a discrepancy, they discuss and reach a consensus. If consensus cannot be achieved, the sample is excluded from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Lei, Study Chair — Fuyong People's Hospital of Bao'an District, Shenzhen
Locations (1):
- Department of Rehabilitation, Fuyong People's Hospital of Bao'an District, Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The Individual Participant Data (IPD) will not be shared due to patient privacy concerns and confidentiality regulations. Protecting sensitive personal and medical information is a priority, and the data contains details that cannot be fully anonymized. Additionally, the data is intended solely for this specific study and is not designed for external distribution or secondary analysis.

REFERENCES:
- [Derived] Song C, Lei B, Li Z, Li H, Tian S, Feng N. Discovery of Posture Secret manual therapy for post-stroke shoulder pain: study protocol for a randomized controlled trial. Front Neurol. 2025 Sep 12;16:1594560. doi: 10.3389/fneur.2025.1594560. eCollection 2025. PMID 41018195